CLINICAL TRIAL: NCT00760721
Title: Increasing Hepatitis B Screening Among Korean Church Attendees (Component Project) Program Project Title: Liver Cancer Control Interventions for Asian Americans
Brief Title: Increasing Hepatitis B Screening Among Korean Church Attendees
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: P01CA109091-01A1 (NIH); P01CA109091-01A1 (NIH)
Record Dates: First submitted 2008-09-25; First posted 2008-09-26 (Estimated); Last update posted 2016-11-28 (Estimated); Status verified 2016-11

CONDITIONS: Hepatitis B
Keywords: Hepatitis B Screening; Korean Americans
MeSH Terms: conditions — Hepatitis B

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Educational small group session with HBV screening resources provided
  Interventions: Behavioral: Educational Small Group Session
- 2 (Sham Comparator): Educational small group discussion, diet/physical activity resources provided
  Interventions: Behavioral: Educational Small Group Session

INTERVENTIONS:
Behavioral: Educational Small Group Session — 1 hour small group health-related discussion

SUMMARY:
The purpose of this study is to design an intervention to increase hepatitis B (HBV) screening among Korean Americans.

The investigators will design a culturally specific intervention (educational sessions) and test the effect of the intervention on 1200 Korean Americans.

All subjects will be interviewed before the intervention/control sessions and 6 months after the sessions to assess HBV screening levels in the two groups. Self-reported HBV screening will be verified by a review of subjects' medical records.

The primary study hypothesis is that the intervention group will have a higher rate of HBV serologic testing at follow-up compared to the control group.

DETAILED DESCRIPTION:
The purpose of this study is to design an intervention to increase hepatitis B (HBV) screening among Korean Americans.

The investigators will design a culturally specific intervention; an educational small group discussion led by a trained Korean leader. The effect of the intervention will be tested on 1200 Korean Americans.

Subjects will be recruited at Korean churches and invited to join a one-hour discussion of health issues with other members of their church. One half of the subjects will participate in the intervention group. These subjects will discuss HBV and will receive resources related to HBV and where to obtain screening. The other half of the subjects will participate in the control group. These subjects will discuss nutrition and physical activity and will receive resources related to these topics, but not related to HBV and where to obtain screening.

All subjects will be interviewed before the sessions and 6 months after the sessions to assess HBV screening levels in the two groups. Self-reported HBV screening will be verified by a review of subjects' medical records.

The primary study hypothesis is that the intervention group will have a higher rate of HBV serologic testing at follow-up compared to the control group.

Secondary hypotheses are:

The intervention group will have a higher level of knowledge of hepatitis B and liver cancer at follow-up compared to the control group.

The effect of the intervention on hepatitis B serologic testing will be mediated by knowledge of hepatitis B and liver cancer.

ELIGIBILITY:
Inclusion Criteria:

* Korean ancestry
* Have not previously received HBV screening or do not know the results of previous HBV screening test
* No history of liver cancer or liver disease
* Current resident of the Los Angeles area

Exclusion Criteria:

* Younger than 18 years of age or Older than 64 years of age
* Not of Korean ancestry
* Previously screened for HBV
* History of liver disease or liver cancer
* Not a current resident of the Los Angeles area

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 1123 (Actual)
Dates: Start 2006-09; Primary Completion 2011-08 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Obtaining HBV Screening Test | 6 months post-intervention

SECONDARY OUTCOMES:
Knowledge and Attitudes Regarding HBV Screening | 6 months post-intervention

CONTACTS AND LOCATIONS:
Overall Officials: Roshan Bastani, PhD, Principal Investigator — University of California, Los Angeles
Locations (1):
- UCLA, Division of Cancer Prevenion and Control Research, Los Angeles, California, United States

REFERENCES:
- [Result] Bastani R, Glenn BA, Maxwell AE, Jo AM, Herrmann AK, Crespi CM, Wong WK, Chang LC, Stewart SL, Nguyen TT, Chen MS Jr, Taylor VM. Cluster-Randomized Trial to Increase Hepatitis B Testing among Koreans in Los Angeles. Cancer Epidemiol Biomarkers Prev. 2015 Sep;24(9):1341-9. doi: 10.1158/1055-9965.EPI-14-1396. Epub 2015 Jun 23. PMID 26104909